CLINICAL TRIAL: NCT00435747
Title: A Double-Blind Comparative Multicenter Study Of The Efficacy And Safety Of Parecoxib IV/IM 40 Mg Vs Placebo On Reducing Opioids Consumption Following Sub Muscular Breast Augmentation Surgery
Brief Title: Efficacy And Safety Of Parecoxib IV/IM 40 Mg Vs Placebo Following Sub Muscular Breast Augmentation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3481100
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib

INTERVENTIONS:
Drug: PARECOXIB SODIUM

SUMMARY:
The present study aims to compare the pre-emptive analgesic efficacy of parecoxib 40 mg IV/IM versus placebo on reducing postoperative acute pain following submuscular breast augmentation. Additionally this study is being conducted to evaluate the safety and tolerability of parecoxib in this kind of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of any ethnic origin aged 18 years or over.
* The patient is post-menopausal, surgically sterile, or using adequate contraception, not lactating, with a negative urine pregnancy test at screening, prior to administration of study medication.
* The patient's preoperative health is graded as a class I or II according to the ASA physical status classification and on the basis of medical history and physical examination.

Exclusion Criteria:

* The patient has significant clinical signs and symptoms suggestive of renal or hepatic morbid conditions
* The patient has a history of clinically significant hypersensitivity to any NSAIDs, cyclooxygenase inhibitors, analgesics or sulfa medications which has a cross sensitivity to the medications used in this study.
* The patient used analgesics or other agents (antidepressants, sedating antihistamines or other sedatives, muscle relaxants, narcotics, or corticosteroids) during the four hours preceding the procedure that could confound the analgesic responses.
* Subjects with a history of established ischemic heart disease (e.g. myocardial infarction, stable angina, unstable angina), peripheral arterial disease and/or cerebrovascular disease (e.g. ischemic or hemorrhagic stroke, transient ischemic attack), as well as subjects with previous revascularization procedure to coronary, carotid, cerebral, renal, aortic or peripheral arterial vasculature

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To evaluate the opioid-sparing effect of parecoxib 40 mg IV/IM compared to placebo in pre emptive analgesia in patients submitted to sub muscular breast augmentation during the first 24 hours after the first dose of study drug.

SECONDARY OUTCOMES:
To evaluate the efficacy, safety and tolerability of parecoxib 40 mg IV/IM compared to placebo used to reduce pain following sub muscular breast augmentation in terms of pain intensity
To evaluate the efficacy, safety and tolerability of parecoxib 40 mg IV/IM compared to placebo used to reduce pain following sub muscular breast augmentation in terms of global evaluation of study medication
To evaluate the efficacy, safety and tolerability of parecoxib 40 mg IV/IM compared to placebo used to reduce pain following sub muscular breast augmentation in terms of vital signs
To evaluate the efficacy, safety and tolerability of parecoxib 40 mg IV/IM compared to placebo used to reduce pain following sub muscular breast augmentation in terms of coagulation tests
To evaluate the efficacy, safety and tolerability of parecoxib 40 mg IV/IM compared to placebo used to reduce pain following sub muscular breast augmentation in terms of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3481100&StudyName=Efficacy%20And%20Safety%20Of%20Parecoxib%20IV/IM%2040%20Mg%20Vs%20Placebo%20Following%20Sub%20Muscular%20Breast%20Augmentation